CLINICAL TRIAL: NCT06762756
Title: What is the Effect of Presenting Evidence of the Mental Vs Physical Health Benefits of Quitting Smoking on Motivation to Stop Smoking? an Online Randomised Controlled Experiment
Brief Title: Impact of Positive Mental Vs. Physical Health Messaging on Motivation to Stop Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katherine Sawyer (Other)
Responsible Party: Sponsor-Investigator, Katherine Sawyer, PhD Student, University of Bath
Organization: University of Bath (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-244
Record Dates: First submitted 2024-12-19; First posted 2025-01-08 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Smoking, Tobacco
Keywords: Smoking; Smoking cessation; Public health; Mental health; Tobacco warning labels
MeSH Terms: conditions — Tobacco Smoking; Smoking; Smoking Cessation; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The intervention was tobacco warning labels with three conditions: i) positive mental health labels; ii) positive physical health labels; iii) blank labels. Participants were randomly allocated to one label condition using Qualtrics embedded randomisation function, stratified by mental health status, and viewed four labels for at least 10 seconds each.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Positive mental health labels (Experimental): Participants viewed four messages, formatted as tobacco packaging labels, communicating the benefits of smoking cessation for mental health. The messages were:
  * "Quitting smoking improves your mental health"
  * "Quitting smoking reduces feelings of depression"
  * "Quitting smoking reduces feelings of anxiety"
  * "Quitting smoking can improve your mood"
  Interventions: Behavioral: Messages on tobacco packaging labels
- Positive physical health labels (Active Comparator): Participants viewed four messages, formatted as tobacco packaging labels, communicating the benefits of smoking cessation for physical health. The messages were:
  * "Quitting smoking improves your health"
  * "Quitting smoking reduces risk your risk of having a heart attack"
  * "Quitting smoking reduces shortness of breath and coughing"
  * "Quitting smoking can improve your oral health"
  Interventions: Behavioral: Messages on tobacco packaging labels
- Blank labels (Placebo Comparator): Participants viewed four blank messages, formatted as tobacco packaging labels. The messages were:
  * Blank template
  * Template with "Example"
  * Template with "Template"
  * Template with "Image, Text"
  Interventions: Behavioral: Messages on tobacco packaging labels

INTERVENTIONS:
Behavioral: Messages on tobacco packaging labels — The intervention was messages of the benefits of smoking cessation formatted as tobacco packaging labels with three conditions. Participants viewed the messages online. There were four messages in each condition. The intervention was informed by relevant patient and public groups.

SUMMARY:
This study tested whether positive messages on tobacco packaging about the mental health benefits of quitting smoking could help motivate people to stop smoking. It compared three types of labels: ones focusing on mental health benefits, ones focusing on physical health benefits, and blank labels.

The experiment involved 631 people who smoke who were randomly shown one of these label types on an online survey platform. Participants' motivation to quit smoking was measured before and after viewing the labels.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported weekly tobacco smokers
2. Aged at least 18 years
3. Could read English

Exclusion Criteria:

Did not smoke tobacco at least weekly

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Motivation to stop smoking | At baseline and follow up immediately after viewing the labels
  Motivation to stop smoking was measured using the Motivation to Stop Scale (MTSS). The MTSS asks participants "Which of the following best describes you?" with the following ordinal scale: 1) "I don't want to stop smoking"; 2) "I think I should stop smoking but don't really want to"; 3) "I want to stop smoking but haven't thought about when"; 4) "I REALLY want to stop smoking but I don't know when I will"; 5) "I want to stop smoking and hope to soon"; 6) "I REALLY want to stop smoking and intend to in the next 3 months"; 7) "I REALLY want to stop smoking and intend to in the next month".

SECONDARY OUTCOMES:
Intention to Quit | Measured at baseline and follow up immediately after viewing the labels
  Participants were asked their intention to quit smoking "Are you planning to quit smoking within the next month?" using a 10-point visual analogue scale, where 1 indicates low intention to quit and 10 indicates higher intention to quit smoking
Quitting Self-Efficacy | Measured at baseline and follow up immediately after viewing the labels
  To measure participants' self-efficacy to quit smoking, participants responded to the questions "Overall, how confident are you that you can stop smoking within the next month?" on a 5-point scale 1 ('not at all') to 5 ('completely confident') and "For me cutting down on the number of cigarettes that I smoke in the next month would be…." On a scale off 1 ('very difficult') to 5 ('very easy'). The mean score across the two items was calculated, with a higher score indicating higher self-efficacy
Smoking Beliefs | Measured at baseline and follow up immediately after viewing the labels
  Participants rated their agreement to the statements "smoking helps people relax", "smoking helps to reduce stress", "smoking helps to keep weight down" "smoking increases social comfort" "those who smoke are more popular" and "second hand smoke is not harmful" using a 5-point scale from 1 ('not at all') to 5 ('a lot'). The mean score across the five items was calculated, with a higher score indicating more favourable beliefs towards smoking
Attention | Measured at follow up immediately after viewing the labels
  Participants rated two statements 'these labels are worth remembering' and 'these labels grabbed my attention' on a 5-point scale from 1 ('not at all') to 5 ('a lot'), mean score across the two items was calculated, with a higher score indicating greater attention
Affective Reactions | Measured at follow up immediately after viewing the labels
  To measure affective reactions to the health labels we used the Self-Assessment Manakin (SAM, (Bradley & Lang, 1994)). Participants rated their affective reactions: valence, arousal, and dominance on a 9-point visual analogue scale. Scales for valence range from 1 'unpleasant' to 9 'pleasant', arousal ranged from 1 'calm' to 9 'excited', and dominance ranged from 1 'controlled' to 9 'in control' with 5 as neutral for all items
Believability | Measured at follow up immediately after viewing the labels
  Perceptions of believability of the health label were measured using the question "How believable are these health labels?", participants rated this on a 5-point scale from 1 ('not at all') to 5 ('a lot')

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Taylor, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analysed during the current study are available in the University of Bath repository.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be available on publication and indefinitely
Access Criteria: Scripts are available at https://osf.io/v5deq/?view_only=d5dd1f5903a0480d94402c7c6528c6a4

REFERENCES:
- [Derived] Sawyer K, Hanafi A, Freeman TP, Burke C, Adams S, Aveyard P, Jacobsen P, Taylor G. What is the effect of presenting evidence of the mental vs physical health benefits of quitting smoking on motivation to stop smoking? An online randomised controlled experiment. BMC Public Health. 2025 Jul 3;25(1):2331. doi: 10.1186/s12889-025-22795-0. PMID 40610984
- See also: Pre-registered protocol on Open Science Framework — https://doi.org/10.17605/OSF.IO/3C75J
- Available data/document: Individual Participant Data Set — https://researchdata.bath.ac.uk — The datasets generated and/or analysed during the current study are available in the University of Bath repository.
- Available data/document: Analytic Code — https://osf.io/v5deq/?view_only=d5dd1f5903a0480d94402c7c6528c6a4 — Scripts are available on Open Science Framework